CLINICAL TRIAL: NCT05830409
Title: Effect of Multisensory Stimulation on Pain During the Preterm Infant's Eye Examination
Brief Title: Multisensory Stimulation in Infants for Eye Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Tasdemir, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MAKU23-1
Record Dates: First submitted 2023-03-29; First posted 2023-04-26 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Premature Retinopathy; Pain, Eye
Keywords: preterm infants; Multisensorial stimulation
MeSH Terms: conditions — Retinopathy of Prematurity; Eye Pain

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisensorial Stimulation Group (Experimental): Preterm newborns who will receive multisensory stimulation during the eye examination.
  Interventions: Behavioral: Multisensorial Stimulation
- Control Group (No Intervention): Preterm newborns who will receive routine care during the eye examination

INTERVENTIONS:
Behavioral: Multisensorial Stimulation — Strategies such as touching, calling, making sense of smell, entering the eye area, and activating the sense of taste will be applied to activate the five senses of the newborn.
  Arms: Multisensorial Stimulation Group

SUMMARY:
This study aimed to evaluate the effects of multisensory stimulation on pain and physiological parameters resulting from ROP examination in preterm newborns.

It was planned as a randomized controlled trial. trying to reach 80 newborns in total. Multisensory stimulation will be applied to the intervention group during the examination. In the control group, routine care will be applied during the examination.

DETAILED DESCRIPTION:
Preterm retinopathy may develop due to intubation in preterm newborns. Therefore, this population undergoes eye examinations at regular intervals. This procedure is painful procedure for babies. Nurses can apply interventions to reduce this pain. In this study, it was planned to apply multisensory stimulation to reduce the pain of the newborn. A randomized controlled trial and routine care were planned in the control group. Neonatal pain will be assessed using the PIPP scale.

ELIGIBILITY:
Inclusion Criteria:

* According to the registry, premature neonates with a gestational age of ≤ 32 weeks or newborns with a birth weight of < 1500 g.
* Newborns undergoing a first-time eye exam to screen for retinopathy of prematurity.

Exclusion Criteria:

* Newborns who need CPR during the examination.
* Newborns experience apnea during the examination.

Ages: 32 Weeks to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Newborns younger than 36 weeks of gestational age
Enrollment: 80 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Pain level | first 30 minutes during procedure
  Premature Infant Pain Profile (PIPP) to be used to assess newborn pain.

SECONDARY OUTCOMES:
Heart rate | first 30 minutes during procedure
  defines the newborn's heart rates per minutes.
Oksigen saturation | first 30 minutes during procedure
  defines the newborn's Oksigen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Halil I Taşdemir, PhD, Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
will be decided later